CLINICAL TRIAL: NCT02787044
Title: INfluenza Vaccine to Effectively Stop Cardio Thoracic Events and Decompensated Heart Failure
Acronym: INVESTED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Wisconsin, Madison (Other); University of Toronto (Other); Boston VA Research Institute, Inc. (Other); Patient-Centered Outcomes Research Institute (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Scott David Solomon, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015P001823; U01HL130163 (NIH)
Record Dates: First submitted 2016-05-25; First posted 2016-06-01 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: influenza vaccine; cardiopulmonary hospitalization; heart failure; myocardial infarction; clinical trial
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Influenza Vaccine (Experimental): High Dose Influenza Vaccine
  Interventions: Biological: High Dose Trivalent Influenza Vaccine
- Standard Dose Influenza Vaccine (Active Comparator): Standard Dose Influenza Vaccine
  Interventions: Biological: Standard Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: High Dose Trivalent Influenza Vaccine — High Dose Trivalent Influenza Vaccine
  Arms: High Dose Influenza Vaccine
Biological: Standard Dose Quadrivalent Influenza Vaccine — Standard Dose Quadrivalent Influenza Vaccine
  Arms: Standard Dose Influenza Vaccine

SUMMARY:
INVESTED will test the hypothesis that high dose trivalent influenza vaccine will reduce cardiopulmonary events to a greater extent than standard dose quadrivalent influenza vaccine in high-risk cardiovascular patients with a recent history of myocardial infarction or heart failure. The trial will enroll 9300 participants over one Vanguard (pilot) season and three additional influenza seasons. The primary endpoint will be a composite of all-cause mortality or cardiopulmonary hospitalization.

DETAILED DESCRIPTION:
Influenza leads to significant morbidity and mortality, particularly in patients with cardiovascular disease. Influenza-related death is more common in patients with cardiovascular disease than any other chronic health condition. Influenza infection has been temporally associated with acute cardiovascular events, such as acute coronary syndrome and acute heart failure. Due to the increased risk for influenza-related complications, annual influenza immunization is recommended by the Centers for Disease Control and Prevention, (CDC) the American Heart Association, and the American College of Cardiology, and widespread influenza vaccination has been associated with reduced cardiac-related hospital admissions, acute exacerbations of heart failure, and winter mortality. Moreover, a meta-analysis has shown that annual vaccination reduces the risk for major adverse cardiovascular events (MACE) by 36%, with a more prominent effect in those with recent acute myocardial infarction (AMI).

Several lines of evidence suggest that a strategy of utilizing high-dose influenza vaccine in at risk cardiovascular patients would reduce morbidity and mortality. Immune responses to influenza vaccine, normally subject to variability by age and concomitant medical conditions, are substantially reduced in patients with heart failure evidenced by lower vaccine-induced antibody titers compared to healthy controls. In a randomized trial, antibody responses in patients with heart failure were augmented by using a higher dose of influenza vaccine. In a meta-analysis, higher dose influenza vaccination was associated with a 27% reduced risk for MACE compared to standard dose vaccine. A randomized study of high dose versus standard dose influenza vaccine in medically-stable patients over age 65 showed that participants receiving high dose vaccine had a 24% reduced risk of laboratory-confirmed influenza associated with protocol-defined influenza-like-illness, and had a low risk for adverse events. High dose influenza vaccine is FDA approved for use in medically stable adults over the age of 65, but has not been studied for patients under the age of 65 or in those with unstable, high risk medical conditions. The CDC does not preferentially recommend one influenza vaccine over another, and the optimal vaccine formulation that offers the most clinical protection in these high risk patients is unknown.

The high morbidity and health care costs among patients with high risk cardiovascular disease along with the reduced immune responses to standard dose influenza vaccines in patients with heart failure provides a compelling rationale to investigate alternative influenza vaccination strategies in this group. INVESTED is an outcomes study in patients with recent acute myocardial infarction (AMI) or heart failure (HF) to test whether a four-fold higher dose of trivalent influenza vaccine will reduce morbidity and mortality compared to standard dose quadrivalent vaccine. INVESTED will test the hypothesize that high dose vaccine will reduce the composite of all cause death or cardiopulmonary hospitalizations in this population, with the following specific aims:

Specific Aim 1. To test the hypothesis that high dose trivalent influenza vaccine will reduce the composite of death or cardiopulmonary events compared with standard dose quadrivalent influenza vaccine in high-risk cardiovascular patients. Patients with recent AMI or HF hospitalization will be randomized to high dose versus standard dose vaccine for up to three influenza seasons. The primary endpoint will be time to first occurrence of death or cardiopulmonary hospitalization within each influenza season. Hospitalizations will be ascertained utilizing multiple approaches (phone, patient report, and electronic health records). Key secondary outcome measures will include total (first and recurrent) cardiopulmonary hospitalizations or death, time to first occurrence of cardiovascular death or cardiopulmonary hospitalization, time to occurrence of all-cause death or cardiopulmonary hospitalization across all enrolled influenza seasons, time to occurrence of all-cause death, and time to first occurrence of cardiopulmonary hospitalizations.

Specific Aim 2. To test the hypothesis that antibody titers to influenza vaccine antigens are associated with cardiopulmonary outcomes. In a subset of participants, antibody titers by hemagglutination inhibition assays to influenza vaccine antigens at baseline and at 4 weeks following randomization will be determined, corresponding to achievement of maximal antibody titer levels after vaccination. The association between geometric mean titers post-vaccination and the occurrence of death or cardiopulmonary hospitalization (primary outcome measure of Specific Aim 1) will be assessed.

Other key correlative study (immune) outcome measures will include:

Change in antibody titers at 4 weeks post-vaccination from baseline to influenza vaccine antigens Seroconversion (demonstration of 4-fold rise in antibody concentrations from baseline) and seroprotection (demonstration of antibody titer level of 1:40) to A/H1N1, A/H3N2, and B-type vaccine antigens

The results of this trial have the potential to inform health care policy regarding optimal influenza vaccination for individuals with high risk cardiovascular disease, which may in turn reduce morbidity from this annual threat to health stability in patients with cardiovascular conditions.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* history of hospitalization for myocardial infarction within 1 year of enrollment OR a history of hospitalization for heart failure within 2 years of enrollment
* At least one of the following additional risk factors:

  * Prior MI (if HF the index event above; or a second MI)
  * Prior HF hospitalization (if MI the index event above; or a second HF event)
  * Age ≥ 65
  * Left ventricular ejection fraction (LVEF) < 40%
  * Diabetes mellitus
  * Obesity (BMI ≥ 30)
  * Renal impairment (eGFR ≤ 60)
  * History of ischemic stroke
  * History of peripheral artery disease
  * Current smoking

Exclusion Criteria:

* Known allergy, hypersensitivity (anaphylaxis), or Guillain-Barré Syndrome within 6 weeks after influenza vaccine
* Any non-cardiac condition that in the opinion of the investigator would lead to life expectancy less than 9 months.
* Receipt of influenza vaccine during current influenza season
* Any illness requiring treatment with antibiotics or anti-inflammatory medication within the past 14 days.
* Any fever over 100 degrees Fahrenheit or 38 degrees Celsius within the past 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5388 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orly Vardeny, PharmD, MS, Principal Investigator — University of Minnesota; Scott D Solomon, MD, Principal Investigator — Brigham and Women's Hospital; KyungMann Kim, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (190):
- United States (127):
  - Birmingham VAMC, Birmingham, Alabama
  - University of Alabama Hypertension Program, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Alaska Heart & Vascular Institute, Anchorage, Alaska
  - Banner University Medicine North, Tucson, Arizona
  - University of Arizona- Sarver Heart Center, Tucson, Arizona
  - CAVHS, Little Rock, Arkansas
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Long Beach VAMC, Long Beach, California
  - University of California Davis Medical Center, Sacramento, California
  - VA San Diego Healthcare System, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - VA West Haven, West Haven, Connecticut
  - Washington DC VAMC, Washington D.C., District of Columbia
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - N FL/S GA Veterans Health System, Gainesville, Florida
  - OneFlorida CDRN, Gainesville, Florida
  - Clearwater Cardiovascular Consultants-Largo, Largo, Florida
  - Inpatient Research Corporation, Miami, Florida
  - ITB Research, Miami, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Clearwater Cardiovascular Consultants-SH, Safety Harbor, Florida
  - Bond Community Health Center, Inc., Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Atlanta VA Health Care System, Decatur, Georgia
  - Peidmont Fayette, Fayetteville, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Chicago Medical Research, Hazel Crest, Illinois
  - Northwester Medicine Lake Forest, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - UnityPoint Health Methodist, Peoria, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - St. Vincent Medical Group, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - VA Eastern Kansas Health Care System, Leavenworth, Kansas
  - Robley Rex VA, Louisville, Kentucky
  - The Heart Clinic of Hamond, Hammond, Louisiana
  - Southeast Louisiana Veterans Healthcare System, New Orleans, Louisiana
  - Ochsner Health System- Baton Rouge, New Orleans, Louisiana
  - ENRM VA Hospital, Bedford, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Charles River Medical Associates, Natick, Massachusetts
  - Boston/West Roxbury VA Hospital, West Roxbury, Massachusetts
  - VA Boston Healthcase System, West Roxbury, Massachusetts
  - VA Ann Harbor Healthcare System, Ann Arbor, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - HealthPartners - Riverside Research, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - VA St. Louis Health Care System, St Louis, Missouri
  - St. Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Heart Institute- Grand Island, Grand Island, Nebraska
  - Darthmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cardio Assoc. of the Del. Valley- Elmer, Elmer, New Jersey
  - Cardio. Assoc. of the Del. Valley- Haddon Heights, Haddon Heights, New Jersey
  - Cardio. Assoc. of the Del. Valley- Sewell, Sewell, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - New Mexico VA Health Care System, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian Queens Bayside/Whitestone, Flushing, New York
  - New York Presbyterian/Queens, Flushing, New York
  - NYPQ - Cardiology Outpatient Clinic, Flushing, New York
  - Winthrop University Hospital, Mineola, New York
  - New York VA, New York, New York
  - NYU Langone Medical Center, New York, New York
  - New York Presbyterian, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Charles George VA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke, Durham, North Carolina
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Heart House Research Foundation, Springfield, Ohio
  - Oregon Health & Science, Portland, Oregon
  - VA Portland Health Care Systems (VAPHCS), Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Providence VA Medical Center, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - WJB Dorn VAMC, Columbia, South Carolina
  - Palmetto Research Center, LLC, Spartanburg, South Carolina
  - VAMC Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Tennessee Valley Healthcare Systems-Nashville, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Austin Heart- Heart Hospital, Austin, Texas
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - Michael E. DeBakey VAMC, Houston, Houston, Texas
  - Houston Heart & Vascular Associates, Kingwood, Texas
  - Houston Methodist Research Institute-CCAT Pearland, Pearland, Texas
  - St. David's Heath & Vascular PLLC, Round Rock, Texas
  - South Texas Veterans Healthcare System, San Antonio, Texas
  - STAR Clinical Trials, San Antonio, Texas
  - Austin Heart San Marcos, San Marcos, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - University of Utah, Salt Lake City, Utah
  - George E. Wahlen Dept of VA Affairs Medical Center, Salt Lake City, Utah
  - VA Medical Center White River Junction, White River Junction, Vermont
  - Inova Heart and Vascular Institute, Alexandria, Virginia
  - Carient Heart & Vascular, Manassas, Virginia
  - Louis A Johnson VAMC, Clarksburg, West Virginia
  - Gundersen Clinic, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - Willam S. Middleton Memorial Veterans Hospital, Madison, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Research Institute, LLC, Milwaukee, Wisconsin
  - Celement J. Zablocki VA Medical Center, Milwaukee, Wisconsin
- Canada (62):
  - TotalCardiology, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - CK Hui Heart Centre, Royal Alexandra Hospital, Edmonton, Alberta
  - Dr. MPJ Senaratne Professional Corporation, Edmonton, Alberta
  - Northwest Echocardiolography, Grande Prairie, Alberta
  - The CARe Clinic (Central Alberta Research), Red Deer, Alberta
  - University of Alberta Hospital- Mazankoski Heart Institute, Edmonton, British Columbia
  - Kelowna General Hospital, Kelowna, British Columbia
  - SMH Cardiology Clinical, Surrey, British Columbia
  - Manna Research Inc. (Vancouver), Vancouver, British Columbia
  - Vancouver General Hospital - Gordon Leslie Diamond Centre, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface Hospital/University of Manitoba, Winnipeg, Manitoba
  - University of Sherbrooke, Dieppe, New Brunswick
  - G.A Research Associates Ltd., Moncton, New Brunswick
  - QEII Health Sciences, Halifax, Nova Scotia
  - Brampton Research Assocaites, Brampton, Ontario
  - Manna Research Inc. (Burlington North), Burlington, Ontario
  - Manna Research Inc. (Burlington South), Burlington, Ontario
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - Vizel Cardiac Research, Cambridge, Ontario
  - Dr. Alan David Bell, Downsview, Ontario
  - Health Sciences North Research Institute, Greater Sudbury, Ontario
  - Dr. D. Shukla Professional Medicine Corporation, Greater Sudbury, Ontario
  - Dr. R. Labonte Professional Medicine Corporation, Greater Sudbury, Ontario
  - Hamilton Health Sciences General Hospital/ McMaste, Hamilton, Ontario
  - Queen's University CardioPulmonary Unit, Kingston, Ontario
  - St. Joseph's Health Care, London, Ontario
  - Dixie Medical Group, Mississauga, Ontario
  - Apple Hills Medical Associates, Mississauga, Ontario
  - PACE, Newmarket, Ontario
  - North York General Hospital, North York, Ontario
  - Sewa Ram Singal Med Prof Corporation, North York, Ontario
  - Heart Care Research, Oshawa, Ontario
  - Dr. James Cha, Oshawa, Ontario
  - Montfort Hospital and Ottawa Cardiovascular Centre, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Heart Function Clinic Queensway Carleton, Ottawa, Ontario
  - Kawartha Cardiology, Peterborough, Ontario
  - St. Catherines Hospital, Saint Catherines, Ontario
  - Scarborough General Hospital, Scarborough Village, Ontario
  - Manna Research (Stoney Creek), Stoney Creek, Ontario
  - Thunder Bay Regional Health Sciences Center, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
  - iHealthCentre, Vaughan, Ontario
  - CISSS de Laval, Hopital Cite de la Sante, Laval, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CIUSSS NÎM Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Manna Research Inc. (Montreal), Montreal, Quebec
  - IUCPQ, Québec, Quebec
  - Centre hospitalier régional de Lanaudière, Saint-Charles-Borromée, Quebec
  - CISSSI- Hopital Pierre-Le Gardeur, Terrebonne, Quebec
  - Centre Hospitalier de Regional Trois-Rivieres, Trois-Rivières, Quebec
  - Prairie Vascular Research Inc., Regina, Saskatchewan
- VA Caribbean Healthcare System, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to NIH data sharing rules
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available as per NIH guidelines on December 4, 2022 (2 years from the primary study publication date).
Access Criteria: Data will be available to all qualified researchers based on the NIH BIOLINCC criteria.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Vardeny O, Sweitzer NK, Detry MA, Moran JM, Johnson MR, Hayney MS. Decreased immune responses to influenza vaccination in patients with heart failure. J Card Fail. 2009 May;15(4):368-73. doi: 10.1016/j.cardfail.2008.11.009. Epub 2008 Dec 18. PMID 19398087
- [Background] Vardeny O, Moran JJ, Sweitzer NK, Johnson MR, Hayney MS. Decreased T-cell responses to influenza vaccination in patients with heart failure. Pharmacotherapy. 2010 Jan;30(1):10-6. doi: 10.1592/phco.30.1.10. PMID 20030468
- [Background] Van Ermen A, Hermanson MP, Moran JM, Sweitzer NK, Johnson MR, Vardeny O. Double dose vs. standard dose influenza vaccination in patients with heart failure: a pilot study. Eur J Heart Fail. 2013 May;15(5):560-4. doi: 10.1093/eurjhf/hfs207. Epub 2013 Jan 4. PMID 23291729
- [Background] Albrecht CM, Sweitzer NK, Johnson MR, Vardeny O. Lack of persistence of influenza vaccine antibody titers in patients with heart failure. J Card Fail. 2014 Feb;20(2):105-9. doi: 10.1016/j.cardfail.2013.12.008. Epub 2013 Dec 19. PMID 24361852
- [Background] Udell JA, Farkouh ME, Solomon SD, Vardeny O. Does influenza vaccination influence cardiovascular complications? Expert Rev Cardiovasc Ther. 2015 Jun;13(6):593-6. doi: 10.1586/14779072.2015.1044439. Epub 2015 May 14. PMID 25971953
- [Background] Vardeny O, Claggett B, Udell JA, Packer M, Zile M, Rouleau J, Swedberg K, Desai AS, Lefkowitz M, Shi V, McMurray JJV, Solomon SD; PARADIGM-HF Investigators. Influenza Vaccination in Patients With Chronic Heart Failure: The PARADIGM-HF Trial. JACC Heart Fail. 2016 Feb;4(2):152-158. doi: 10.1016/j.jchf.2015.10.012. Epub 2015 Dec 30. PMID 26746371
- [Background] Udell JA, Zawi R, Bhatt DL, Keshtkar-Jahromi M, Gaughran F, Phrommintikul A, Ciszewski A, Vakili H, Hoffman EB, Farkouh ME, Cannon CP. Association between influenza vaccination and cardiovascular outcomes in high-risk patients: a meta-analysis. JAMA. 2013 Oct 23;310(16):1711-20. doi: 10.1001/jama.2013.279206. PMID 24150467
- [Background] Vardeny O, Udell JA, Joseph J, Farkouh ME, Hernandez AF, McGeer AJ, Talbot HK, Bhatt DL, Cannon CP, Goodman SG, Anand I, DeMets DL, Temte J, Wittes J, Nichol K, Yancy CW, Gaziano JM, Cooper LS, Kim K, Solomon SD. High-dose influenza vaccine to reduce clinical outcomes in high-risk cardiovascular patients: Rationale and design of the INVESTED trial. Am Heart J. 2018 Aug;202:97-103. doi: 10.1016/j.ahj.2018.05.007. Epub 2018 May 23. PMID 29909156
- [Result] Vardeny O, Kim K, Udell JA, Joseph J, Desai AS, Farkouh ME, Hegde SM, Hernandez AF, McGeer A, Talbot HK, Anand I, Bhatt DL, Cannon CP, DeMets D, Gaziano JM, Goodman SG, Nichol K, Tattersall MC, Temte JL, Wittes J, Yancy C, Claggett B, Chen Y, Mao L, Havighurst TC, Cooper LS, Solomon SD; INVESTED Committees and Investigators. Effect of High-Dose Trivalent vs Standard-Dose Quadrivalent Influenza Vaccine on Mortality or Cardiopulmonary Hospitalization in Patients With High-risk Cardiovascular Disease: A Randomized Clinical Trial. JAMA. 2021 Jan 5;325(1):39-49. doi: 10.1001/jama.2020.23649. PMID 33275134
- [Derived] Lassen MCH, Howell N, Claggett BL, Biering-Sorensen T, Vardeny O, Solomon SD, Udell J, Joseph J, Hegde SM. Educational Attainment Level and Risk of Mortality and Cardiopulmonary Outcomes in High-Risk Patients With Cardiovascular Disease: The INVESTED Trial. J Am Heart Assoc. 2025 Jul;14(13):e040221. doi: 10.1161/JAHA.124.040221. Epub 2025 Jun 18. PMID 40530474
- [Derived] Peikert A, Claggett BL, Udell JA, Joseph J, Hegde SM, Kim K, Mao L, Wang T, Havighurst TC, Farkouh ME, Bhatt DL, Tattersall MC, Cooper LS, Solomon SD, Vardeny O. Influenza Vaccine Immune Response in Patients With High-Risk Cardiovascular Disease: A Secondary Analysis of the INVESTED Randomized Clinical Trial. JAMA Cardiol. 2024 Jun 1;9(6):574-581. doi: 10.1001/jamacardio.2024.0468. PMID 38583091
- [Derived] Hegde SM, Claggett BL, Udell JA, Kim K, Joseph J, Farkouh ME, Peikert A, Bhatt AS, Tattersall MC, Bhatt DL, Cooper LS, Solomon SD, Vardeny O. Temporal Association Among Influenza-Like Illness, Cardiovascular Events, and Vaccine Dose in Patients With High-Risk Cardiovascular Disease: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2331284. doi: 10.1001/jamanetworkopen.2023.31284. PMID 37707817
- [Derived] Wang T, Mao L. Stratified proportional win-fractions regression analysis. Stat Med. 2022 Nov 20;41(26):5305-5318. doi: 10.1002/sim.9570. Epub 2022 Sep 14. PMID 36104953
- [Derived] Vardeny O, Hernandez AF, Cohen LW, Franklin A, Baqai M, Palmer S, Bierer BE, Cobb N. Transitioning to the National Institutes of Health single institutional review board model: Piloting the use of the Streamlined, Multi-site, Accelerated Resources for Trials IRB Reliance. Clin Trials. 2019 Jun;16(3):290-296. doi: 10.1177/1740774519832911. Epub 2019 Mar 13. PMID 30866676
- See also: INVESTED Trial Website — http://investedtrial.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5388 patients were consented for the study. Of these, 15 patients were not randomized (decided not to participate prior to randomization). 5373 patients were randomized and a total of 113 patients were excluded from all efficacy analyses prior to database lock because they had been enrolled at a site that was closed for major violations of good clinical practice, leaving 5260 participants in the efficacy and safety analysis.
Period: Overall Study
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine
Started (Total Randomized patients) | 2630 | 2630
Completed | 2615 | 2611
Not Completed | 15 | 19
Not completed — Lost to Follow-up | 15 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine | Total
Number analyzed (Participants) | 2630 | 2630 | 5260
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.6) | 65.5 (12.5) | 65.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Some patients chose intersex or refused to answer
  Participants
    number analyzed (Participants) | 2621 | 2625 | 5246
    Female | 717 | 756 | 1473
    Male | 1904 | 1869 | 3773
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 250 | 267 | 517
  Not Hispanic or Latino | 2349 | 2334 | 4683
  Unknown or Not Reported | 31 | 29 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 32 | 49
  Asian | 81 | 74 | 155
  Native Hawaiian or Other Pacific Islander | 13 | 12 | 25
  Black or African American | 407 | 377 | 784
  White | 2042 | 2061 | 4103
  More than one race | 12 | 14 | 26
  Unknown or Not Reported | 58 | 60 | 118
Region of Enrollment [Number; unit: participants]
  Canada | 838 | 838 | 1676
  United States | 1792 | 1792 | 3584
Ejection Fraction [Mean (Standard Deviation); unit: Percentage] — Population: Measures not available in all patients
  Percentage
    number analyzed (Participants) | 2275 | 2274 | 4549
    (all) | 42.5 (16.1) | 41.9 (16.2) | 42.2 (16.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Not available on all patients
  kg/m^2
    number analyzed (Participants) | 2622 | 2623 | 5245
    (all) | 30.7 (7.2) | 31.0 (7.7) | 30.9 (7.4)
Qualifying Event [Count of Participants; unit: Participants]
  Heart Failure | 1641 | 1648 | 3289
  Myocardial Infarction | 982 | 978 | 1960
Hypertension [Count of Participants; unit: Participants] | 1986 | 2060 | 4046
Dyslipidemia [Count of Participants; unit: Participants] | 1793 | 1823 | 3616
History of Percutaneous Coronary Intervention [Count of Participants; unit: Participants] | 1103 | 1059 | 2162
Atrial Fibrillation [Count of Participants; unit: Participants] | 854 | 871 | 1725
History of Coronary Artery Bypass Graft [Count of Participants; unit: Participants] | 503 | 537 | 1040
History of Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants] | 486 | 520 | 1006
History of Implantable Cardioverter Defibrillator [Count of Participants; unit: Participants] | 463 | 493 | 956
Asthma [Count of Participants; unit: Participants] | 308 | 294 | 602
Statins (MI group) [Count of Participants; unit: Participants] — Population: Reported in MI group only
  Participants
    number analyzed (Participants) | 982 | 978 | 1960
    (all) | 920 | 915 | 1835
Aspirin (MI Group) [Count of Participants; unit: Participants] — Population: Reported in MI group only
  Participants
    number analyzed (Participants) | 982 | 978 | 1960
    (all) | 907 | 878 | 1785
Beta Blocker (MI Group) [Count of Participants; unit: Participants] — Population: Reported in MI group only
  Participants
    number analyzed (Participants) | 982 | 978 | 1960
    (all) | 839 | 840 | 1679
Diuretic (HF group) [Count of Participants; unit: Participants] — Population: Reported in HF group only
  Participants
    number analyzed (Participants) | 1641 | 1648 | 3289
    (all) | 1294 | 1313 | 2607
ACE Inhibitor/ Angiotensin Receptor Blocker / Angiotensin Receptor Neprilysin Inhibitor [Count of Participants; unit: Participants] — ACE = Angiotensin Converting Enzyme Population: Reported in HF group only
  Participants
    number analyzed (Participants) | 1641 | 1648 | 3289
    (all) | 1086 | 1111 | 2197
Mineralocorticoid Receptor Antagonist (MRA) (HF group) [Count of Participants; unit: Participants] — Population: Reported in HF group only
  Participants
    number analyzed (Participants) | 1641 | 1648 | 3289
    (all) | 572 | 546 | 1118
Digoxin (HF Group) [Count of Participants; unit: Participants] — Population: Reporte in HF group only
  Participants
    number analyzed (Participants) | 1641 | 1648 | 3289
    (all) | 155 | 159 | 314
Beta Blocker (HF Group) [Count of Participants; unit: Participants] — Population: Reported in HF group only
  Participants
    number analyzed (Participants) | 1641 | 1648 | 3289
    (all) | 1381 | 1398 | 2779

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Death or Cardiopulmonary Hospitalization Within Each Vaccination Season
Description: Number of patients with first occurrence of death or cardiopulmonary hospitalization within each vaccination season
Time Frame: Up to 1 year from vaccination (repeats seasonally)
Measure: Count of Units; unit: Participant-Seasons
Units Other Than Participants: Participant-Seasons
Groups:
- High Dose Influenza Vaccine: High Dose Influenza Vaccine
  High Dose Trivalent Influenza Vaccine: High Dose Trivalent Influenza Vaccine; Note primary analysis is of participant-seasons (n = 3577)
- Standard Dose Influenza Vaccine: Standard Dose Influenza Vaccine
  Standard Dose Quadrivalent Influenza Vaccine: Standard Dose Quadrivalent Influenza Vaccine; Note primary analysis is of participant-seasons (n = 3577)
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine
Number analyzed (Participants) | 2630 | 2630
Number analyzed (Participant-Seasons) | 3577 | 3577
Participant-Seasons | 975 | 924
Statistical Analysis 1: Comparison: High Dose Influenza Vaccine vs Standard Dose Influenza Vaccine; Note, each participant can be included in the primary analysis up to 3 times (participating seasons); Test type: Superiority; p = 0.21, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.97 to 1.17]

2. Secondary Outcome: Total Cardiopulmonary Hospitalizations or Death
Description: Total (first and recurrent) cardiopulmonary hospitalizations or death
Time Frame: Up to 3 years
Measure: Number; unit: All CP hospitalizations/death
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine
Number analyzed (Participants) | 2630 | 2630
All CP hospitalizations/death | 1857 | 1784
Statistical Analysis 1: Comparison: High Dose Influenza Vaccine vs Standard Dose Influenza Vaccine; Test type: Superiority; p = 0.44, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.94 to 1.15]

3. Secondary Outcome: Cardiovascular Death or Hospitalization Within Each Vaccination Season
Description: Number of patients with first cardiovascular death or cardiovascular hospitalization within each influenza season
Time Frame: Up to one year from vaccination
Measure: Count of Units; unit: Participant-Seasons
Units Other Than Participants: Participant-Seasons
Groups:
- High Dose Influenza Vaccine: High Dose Influenza Vaccine
  High Dose Trivalent Influenza Vaccine: High Dose Trivalent Influenza Vaccine; Note: primary analysis is of participant-seasons (n = 3577)
- Standard Dose Influenza Vaccine: Standard Dose Influenza Vaccine
  Standard Dose Quadrivalent Influenza Vaccine: Standard Dose Quadrivalent Influenza Vaccine; Note: primary analysis is of participant-seasons (n = 3577)
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine
Number analyzed (Participants) | 2630 | 2630
Number analyzed (Participant-Seasons) | 3577 | 3577
Participant-Seasons | 805 | 752
Statistical Analysis 1: Comparison: High Dose Influenza Vaccine vs Standard Dose Influenza Vaccine; Each participant can be analyzed up to three times (seasons); Test type: Superiority; p = 0.16, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [.97 to 1.2]

4. Secondary Outcome: Death or Cardiopulmonary Hospitalization Across Enrolling Seasons
Description: First cardiopulmonary Hospitalization or all-cause death across enrolling seasons
Time Frame: Up to three years
Measure: Number; unit: first CP hospitalization/death
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine
Number analyzed (Participants) | 2630 | 2630
first CP hospitalization/death | 955 | 918
Statistical Analysis 1: Comparison: High Dose Influenza Vaccine vs Standard Dose Influenza Vaccine; Test type: Superiority; p = 0.26, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [.96 to 1.15]

5. Secondary Outcome: All-Cause Mortality
Description: Number of patients with first occurrence of all-cause mortality
Time Frame: Up to 3 years
Measure: Number; unit: All cause deaths
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine
Number analyzed (Participants) | 2630 | 2630
All cause deaths | 223 | 222
Statistical Analysis 1: Comparison: High Dose Influenza Vaccine vs Standard Dose Influenza Vaccine; Test type: Superiority; p = 0.96, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.84 to 1.21]

ADVERSE EVENTS:
Time Frame: 1 week for post-vaccination adverse events; 1-3 years, depending on length of participation for serious adverse events
Description: Post-vaccination AEs were collected via participant self report up to 1 week post vaccination. Potential SAEs during study participation were reviewed by study monitors. For all-cause mortality, the number of patients at risk are the total number of patients randomized who were included in the efficacy analyses: 2630 per group. For all other adverse events, the safety analysis set consists of patients who received study vaccination (2606 in high-dose group and 2604 in standard-dose group).
Arm/Group | High Dose Influenza Vaccine | Standard Dose Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 223/2630 | 222/2630
Serious Adverse Events (participants affected / at risk) | 2/2606 | 4/2604
Other Adverse Events (participants affected / at risk) | 1241/2606 | 1096/2604
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Influenza Vaccine (N=2606) | Standard Dose Influenza Vaccine (N=2604)
Bell's Palsy (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysgusia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Influenza Vaccine (N=2606) | Standard Dose Influenza Vaccine (N=2604)
Pain at injection site (Injury, poisoning and procedural complications) | 788 (932) | 594 (683)
Myalgia (General disorders) | 447 (500) | 391 (423)
Overall Discomfort (General disorders) | 290 (310) | 266 (280)
Headache (General disorders) | 265 (279) | 253 (272)
Swelling (Injury, poisoning and procedural complications) | 179 (198) | 115 (119)
Erythema (Injury, poisoning and procedural complications) | 144 (157) | 150 (157)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02787044/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT02787044/SAP_001.pdf
  • Informed Consent Form (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT02787044/ICF_002.pdf